CLINICAL TRIAL: NCT01709448
Title: Predictive Modeling of Anal Dysplasia Progression in HIV
Brief Title: Modeling Study to Predict Progression of Anal Cancer Pre-cursor Lesions in HIV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: University of Cincinnati (Other); Cincinnati VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jaime Robertson, Assistant Professor, University of Cincinnati
Other Study IDs: 1K23AI080202-01 (NIH); 1K23AI080202-01 (NIH)
Record Dates: First submitted 2012-10-16; First posted 2012-10-18 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Neoplasms, Squamous Cell; Papillomavirus Infections
Keywords: Neoplasms, Squamous Cell; Papillomavirus Infections; HIV
MeSH Terms: conditions — Neoplasms, Squamous Cell; Papillomavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Anal cytology Anal biopsies
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether a model can be created to predict the progression of early anal cancer precursor lesions in HIV using potential predictors such as: HIV treatment history, smoking history, sexual history, human papillomavirus viral load, human papillomavirus protein expression, and cell markers associated with progression of HPV-related lesions.

DETAILED DESCRIPTION:
Persons living with HIV-infection are at greatly increased risk for anal carcinoma and anal intraepithelial neoplasia (AIN). Despite the overall improvement in HIV outcomes, the incidence of anal carcinoma has not decreased with the advent of highly active antiretroviral ther-apy. Further, there is substantial morbidity and mortality associated with anal carcinoma in HIV-infected individuals. For these reasons, it is critically important to develop effective screening and treatment strategies in this population. Anal carcinoma is similar to cervical carcinoma in that they are both associated with infection with human papillomavirus (HPV) and share similar cytologic features of dysplasia. Anal cytology screening is ultimately expected to reduce the incidence of anal carcinoma similar to that seen with cervical cancer after the introduction of cervical Pap screening. Given the high frequency of abnormal cytology in patients with HIV and the need to confirm results by high-resolution anoscopy, however, the implementation of screening programs requires a substantial commitment of clinical resources. The workload and costs involved in following up on abnormal cytology reduce the cost-effectiveness of screening and pose a significant barrier to its widespread integration into routine HIV care. A model for predicting which patients are at greatest risk for progressive of anal dysplasia is needed in order to decrease the need for excessive confirmatory procedures in this population. Without such a model, anal carcinoma screening may remain cost prohibitive for many HIV clinics.

The objective of this study is to develop a predictive model to identify patients who are at greatest risk for progression of anal intraepithelial neoplastic changes. The central hypotheses are: 1) that progression of early HPV-related anal dysplasia is associated with environmental, virological, and host molecular factors and 2) that it is possible to develop a predictive statistical model with a high sensitivity and specificity for predicting disease progression. These hypotheses have been formulated on the basis of strong evidence from studies of HPV-related cervical dysplasia that smoking, HPV E2 expression, HPV E6/E7 protein expression, high-risk HPV type, HPV viral load, p16 expression, p53 expression and Ki67 expression are associated with progressive cervical dysplasia. The rationale for the proposed research is that development of a predictive model will allow clinicians to design more cost-effective screening and follow-up strategies which focus resources on intensively testing only those patients with a significant risk for progression. Further, the models developed will allow clinicians to identify a population of patients who may benefit from early treatment interventions. Finally, information learned from this research may provide information applicable to other HPV-related cancers.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected
* Age > 18 years old
* Abnormal anal screening cytology

Exclusion Criteria:

* Inability to sign informed consent
* Life-threatening illness or other contraindication for high-resolution anoscopy
* anal intraepithelial neoplasia not confirmed by anal biopsy
* history of anal carcinoma
* history of HPV vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2009-01; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
histological diagnosis of high-grade squamous intra-epithelial lesion confirmed by anal biopsy | 12 months, 24 months, 36 months

SECONDARY OUTCOMES:
Regression of lesions defined by normal appearance on anoscopy and normal histology on anal biopsy following previous diagnosis of squamous intraepithelial lesion. | 12 months, 24 months, 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Jaime C Robertson, MD, Principal Investigator — University of Cincinnati
Locations (2):
- United States (2):
  - Cincinnati VA Medical Center, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio

REFERENCES:
- See also: University of Cincinnati - Division of Infectious Diseases — http://intmed.uc.edu/divisions/infectious_diseases/
- See also: Cincinnati VA Medical Center — http://www.cincinnati.va.gov/